CLINICAL TRIAL: NCT00259883
Title: Post-marketing Clinical Study on PAXIL Tablet in Patients With Depression or Depressive Mood - A Study on Combination of PAXIL Tablet and Benzodiazepines
Brief Title: Combination Of PAXIL Tablet And Benzodiazepines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104228
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Mental Disorders
Keywords: depressive episodes; paroxetine; PAXIL; depression; benzodiazepine; combination
MeSH Terms: conditions — Mental Disorders; Depression | interventions — Paroxetine

ARMS (1):
- paroxetine (Experimental): paroxetine 20 to 40mg/day
  Interventions: Drug: paroxetine

INTERVENTIONS:
Drug: paroxetine — 1 or 2 tablets once a day

SUMMARY:
This study was designed to assess the efficacy and safety of combination therapy of PAXIL and benzodiazepine anxiolytics. PAXIL Tablet will be administered to patients with depression or depressive episodes who have received Benzodiazepines for at least 4 weeks, and changes in the symptoms of depression will be evaluated by use of the rate and extent of decrease in Hamilton Rating Scale for Depression (HAM-D).

ELIGIBILITY:
Inclusion criteria:

* Patients with depression or depressive episodes who are diagnosed to have major depressive disorders according to the DSM-IV criteria.
* Patients with 14 or higher points in total scores for Items No.1 - 17 on HAM-D.
* Patients who have continuously received Benzodiazepine anxiolytics.

Exclusion criteria:

* Patients with a strong suicide tendency.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2005-06; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The rate and extent of decrease in Hamilton Rating Scale for Depression (HAM-D) | 8 weeks

SECONDARY OUTCOMES:
The rate and extent of decrease in each item of HAM-D. The rate and extent of decrease of SRQ-D. Percentage of subjects who started tapering Benzodiazepine dose. Success rate in Benzodiazepine tapering Extent increase of SF-8. CGI responder rate. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site